CLINICAL TRIAL: NCT04651543
Title: Is a Follow-up Radiological Study at One Week Necessary in Conservatively Treated Fractures of the Proximal Humerus? Randomized Prospective Study
Brief Title: X-Ray Follow-up in Proximal Humeral Fractures Conservatively Treated
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital del Mar (Other)
Responsible Party: Principal Investigator, Carlos Torrens, Clinical Professor, Hospital del Mar
Other Study IDs: 102020
Record Dates: First submitted 2020-11-26; First posted 2020-12-03 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-03

CONDITIONS: Shoulder Fractures
Keywords: proximal humeral fractures; conservative treatment; outcomes
MeSH Terms: conditions — Shoulder Fractures | interventions — X-Rays

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- no control X-Ray: patients with a proximal humeral fracture without one-week X-Ray control
  Interventions: Other: X-Ray
- one-week X-Ray control: patients with a proximal humeral fracture with one-week X-Ray control
  Interventions: Other: X-Ray

INTERVENTIONS:
Other: X-Ray — X-ray obtained at one-week of the fracture

SUMMARY:
Randomly assign patients with fractures of the proximal humerus to conservative treatment to a group in which a control radiological study will be carried out after a week of evolution of the fracture and to another group in which this control radiology will not be carried out. In the evolutionary controls, it will be determined whether there are differences between the two groups in the final functional result, in the perception of quality of life, and in the number of complications derived from the fracture.

ELIGIBILITY:
Inclusion Criteria:

* patients> 18 yo and < 85 yo
* Fractures of the proximal humerus <3 weeks of evolution.
* fractures treated conservatively.
* No previous pathology of the affected shoulder.

Exclusion Criteria:

* dementia
* impossibility of carrying out a rehabilitation guideline.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with proximal humeral fractures
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Constant Score (0-100 were 100 is the higher outcomes mean better outcomes) | 2 years
  shoulder functional outcome score

CONTACTS AND LOCATIONS:
Locations (1):
- Parc de Salut Mar, Barcelona, Spain